CLINICAL TRIAL: NCT03811652
Title: A Phase 1/1b Multicenter, Open-label, Dose-escalation, and Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Antitumor Activity of MEDI7247 in Patients With Advanced or Metastatic Disease in Selected Solid Tumors
Brief Title: A Multiple Ascending Dose Study of MEDI7247 in Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8540C00002
Record Dates: First submitted 2018-12-21; First posted 2019-01-22 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Non Small Cell Lung Cancer Squamous (NSCLC-Sq); Head and Neck Squamous Cell Carcinoma (HNSCC); Small Cell Lung Cancer (SCLC); Pancreatic Ductal Adenocarcinoma (PDAC); Colorectal Cancer (CRC); Metastatic Castration-resistant Prostate Cancer (mCRPC)
Keywords: Medi7247; non small cell lung cancer; head and neck cancer; small cell lung cancer; colorectal cancer; prostate cancer; pancreatic adenocarcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Small Cell Lung Carcinoma; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- NSCLC-Sq/HNSCC (Experimental): Patients with advanced or metastatic NSCLC-Sq or HNSCC who have recurrence after, or are refractory or intolerant to standard therapy, including at least one prior standard of care regimen (platinum-based for HNSCC). PDL-1 positive patients should have received previous PD-1 or PD-L1 inhibitor where available.
  Interventions: Drug: MEDI7247
- Small Cell Lung Cancer (Experimental): Patients with advanced SCLC who have recurrence after, or are refractory or intolerant to standard therapy, including at least one prior standard of care regimen.
  Interventions: Drug: MEDI7247
- Colorectal Cancer (Experimental): Patients with metastatic adenocarcinoma of the colon or rectum who have received and have progressed, or have documented intolerance, on prior thymidylate synthase inhibitor (eg, 5-fluorouracil (5-FU), capecitabine, raltitrexed, tegafur-uracil (UFT), irinotecan, and oxaliplatin for metastatic disease. If patients progress within 6 months of their last dose of adjuvant therapy this should be considered as a line of therapy in the metastatic setting. Patients with known RAS wildtype tumors must have received and progressed, or have documented intolerance, on anti-EGFR antibody. Patients with microsatellite instability-high or deficient mismatch repair tumors, must have received and progressed, or have documented intolerance on a PD-1 inhibitor, or PD-1 inhibitor plus cytotoxic T-lymphocyte antigen-4 inhibitor treatment where available.
  Interventions: Drug: MEDI7247
- Pancreatic Ductal Adenocarcinoma (Experimental): Patients with unresectable, locally advanced or metastatic PDAC who have recurrence after, or are refractory or intolerant to standard therapy, including at least one prior line of treatment.
  Interventions: Drug: MEDI7247
- Metastatic Castration-Resistant Prostate Cancer (Experimental): Patients with mCRPC who have received prior treatment with abiraterone or enzalutamide, with or without a prior taxane-based chemotherapy in the mCRPC setting.
  Interventions: Drug: MEDI7247
- Other advanced/metastatic target expressing solid tumors (Experimental): Patients with advanced or metastatic solid tumors not defined by other treatment arms who have positive expression of the protein target and have exhausted all approved therapies
  Interventions: Drug: MEDI7247

INTERVENTIONS:
Drug: MEDI7247 — Subjects with advanced solid tumors will enroll into the respective arms to receive Medi7247 IV at prescribed dose and schedule

SUMMARY:
To assess safety and tolerability, describe the dose-limiting toxicities, assess the preliminary antitumor activity, determine the maximum tolerated dose (MTD) or the highest protocol-defined dose (maximum administered dose) in the absence of establishing the MTD, and a recommended dose for further evaluation of MEDI7247 in patients with selected advanced or metastatic solid tumor malignancies that have received at least 1 prior line of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of advanced or metastatic select solid tumors and either progression on or documented intolerance to standard therapies
2. Age ≥ 18 years at the time of screening.
3. Written informed consent and any locally required authorization
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. At least 1 measurable target lesion by CT or MRI per RECIST Version 1.1 (excluding mCRPC)
6. Adequate Liver Function: Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 × ULN (upper limit normal), Albumin > 3 g/dL, and serum total bilirubin (TBL) ≤ 1.5 × ULN; (unless bilirubin rise is due to Gilbert's syndrome, hepatic metastases or of non-hepatic origin, in which case TBL ≤ 3 × ULN is allowed)
7. Creatinine Clearance (CrCL) ≥ 40 mL/min
8. Adequate Hematopoesis: Absolute Neutrophil Count (ANC) ≥ 1,500/μL, Platelets ≥ 100,000/μL, and Hgb ≥ 9 g/dL unassisted by transfusion or growth factor within 14 days of screening
9. Provision of archival or fresh tumor tissue at screening
10. Female patients of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception, and must agree to continue using such precautions for 90 days after the last dose of investigational product.
11. Nonsterilized male patients who are sexually active with a female partner of childbearing potential must use a male condom plus spermicide from 7 days post-screening and for 90 days after receipt of the last dose of investigational product.

Exclusion Criteria:

1. Active central nervous system (CNS) metastases, unless adequately treated and patients have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) and prednisolone 10 mg or less for more than 2 weeks prior to enrollment. For SCLC, a brain MRI scan that was conducted ≤ 28 days from Day 1 is required.
2. Residual toxicity from prior anticancer therapy not resolved to NCI CTCAE v4.03 Grade 1, with the exception of alopecia/vitiligo at the time of first dose of investigational product. For patients previously receiving immunotherapy, toxicities that are unlikely to recover to Grade 1.
3. Royal Marsden Hospital (RMH) prognostic score 2 and 3 at baseline.
4. Treatment with anticancer therapy including chemotherapy, radiation therapy, immunotherapy, biologic, or any investigational therapy within 21 days, or prior palliative radiotherapy within 2 weeks of the first dose of investigational product.

5 Prior treatment with other Pyrrolobenzodiazepine-Antibody Drug Conjugates.

6 History of previous malignancies (except for locally curable cancers) unless a complete remission was achieved at least 3 years prior to study entry AND no additional therapy is required during the study period (except adjuvant hormonal therapy and bisphosphonate).

7. Failure to recover from major surgery or significant traumatic injury within 21 days of first dose of study treatment.

8 History of hepatic sinusoidal obstruction syndrome, also called veno-occlusive disease 9. History of capillary leak syndrome. 10 Blood transfusion within 14 days of study entry except when needed for disease related anemia.

11. New York Heart Association classes III-IV congestive heart failure or serious cardiac arrhythmia requiring treatment, history of myocardial infarction, unstable angina, vascular stent, or coronary artery bypass graft within 6 months of the first dose of investigational product. 12. Active human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infections at the time of screening.

13. Current severe active systemic disease including active concurrent malignancy 14. Pregnancy and/or breastfeeding at time of screening 15. Concurrent enrollment in anther clinical study involving an investigational treatment that is not an extension of another MedImmune study with the same investigational product.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Events | From time of informed consent through 90 days post end of treatment
  To assess the occurrence of adverse events
Occurrence of Serious Adverse Events | From time of informed consent through 90 days post end of treatment
  To assess the occurrence of serious adverse events
Occurrence of Dose Limiting Toxicities | During the evaluation period of 21 days post first dose
  To assess the occurrence of toxicities and abnormal laboratory results that may limit further dose administration
Number of patients with changes in laboratory parameters from baseline | From time of informed consent through 90 days post end of treatment
  To assess serum chemistry, hematology, urinalysis and coagulation parameters
Number of patients with changes in vital signs parameters from baseline | from time of informed consent through 21 days post last dose
  to assess changes in vital signs
Number of patients with changes in electrocardiogram results from baseline | from time of informed consent through 21 days post last dose
  to assess changes in ECG
Percentage of patients with changes in laboratory parameters from baseline | from time of informed consent through 90 days post end of treatment
  to assess changes in serum chemistry, hematology, urinalysis, and coagulation parameters

SECONDARY OUTCOMES:
MEDI7247 maximum observed concentration (Cmax) | From first dose through 90 days post end of treatment
  To characterize MEDI7247 single agent Pharmacokinetics
MEDI7247 terminal half life (t1/2) | From first dose through 90 days post end of treatment
  To characterize single agent MEDI7247 pharmacokinetics
MEDI7247 area under the concentration/time curve (AUC) | from first dose through 90 days post end of treatment
  To characterize single agent MEDI7247 pharmacokinetics
MEDI7247 clearance | from first dose through 90 days post end of treatment
  to characterize the single agent MEDI7247 pharmacokinetics
Number of subjects who develop anti-drug antibodies | first dose through 90 days post end of treatment
  To characterize MEDI7247 immunogenicity
Best Overall Response | From time of informed consent and up to 90 days post end of treatment
  To assess antitumor activity of MEDI7247
Objective Response Rate (ORR) | From time of informed consent and up to 2 years after last subject in
  To assess antitumor activity of MEDI7247
Time to Response (TTR) | From time of informed consent and up to 90 days post end of treatment
  To assess antitumor activity of MEDI7247
Duration of Response (DoR) | From time of informed consent and up to 2 years after last subject in
  To assess antitumor activity of MEDI7247
Progression Free Survival (PFS) | From time of informed consent and up to 2 years after last subject in
  To assess the antitumor activity of MEDI7247
Disease Control (DC) | From time of informed consent and up to 2 years after last subject in
  To assess antitumor activity of MEDI7247
Overall Survival (OS) | From time of informed consent and up to 2 years after last subject in
  To assess antitumor activity of MEDI7247

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Research Site, Huntersville, North Carolina
  - Research Site, Nashville, Tennessee
- Research Site, Toronto, Ontario, Canada